CLINICAL TRIAL: NCT04730193
Title: The Effect of Caffeine on Cerebrovascular and Retinal Microvessel Reactivity
Brief Title: Caffeine and Cerebrovascular Reactivity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 12731
Record Dates: First submitted 2021-01-19; First posted 2021-01-29 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Caffeine
Keywords: caffeine; Cerebrovascular reactivity; Retinal reactivity
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: subject will take drug A on first session and measurements will be performed at baseline and 1 hour after treatment; subject will come for second visit in 5-7 days and take drug B, measurements will be performed at baseline and 1 hour after treatment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigator, and outcomes assessors are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants randomized to placebo group will receive placebo capsule
  Interventions: Drug: Placebo
- Caffeine (Experimental): Participants randomized to caffeine group will receive 100mg caffeine capsule
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Caffeine, also known as Trimethylxanthine, will be purchased through the University of Oklahoma Health Sciences Pharmacy and formulated into capsule pills containing 100mg of active ingredient
  Other Names: Trimethylxanthine
  Arms: Caffeine
Drug: Placebo — Placebo pill will be formulated with a non active ingredient such as rice flour powder
  Arms: Control

SUMMARY:
Caffeine is the most commonly used stimulant drug with well documented effects on cerebral vascula-ture. Caffeine is known to non-specifically bind to adenosine receptors in the brain and to reduce resting blood flow while improving attention and cognitive function, which suggests that it may allow a more efficient dynamic blood flow regulation through neurovascular coupling. This study will use standardized dose of caffeine to test its effect on NVC responses in cerebral and retinal arterioles.

DETAILED DESCRIPTION:
Normal brain function is critically dependent on moment-to-moment adjustment of cerebral blood flow to match demands of activated neurons. This process is known as neurovascular coupling (NVC) and recent in vivo studies demonstrate that impairment of NVC responses is associated with worse cognitive performance. Several methods are available to measure NVC responses in human subjects, including transcranial Doppler (TCD), functional near infrared spectroscopy (fNIRS), and dynamic retinal vessel analysis (DVA). Although all these methodologies aim to measure hemodynamic changes in the brain vasculature in response to cognitive, motor, or visual stimulation, the responses are evaluated on the different levels of cerebral vasculature including microvasculature (fNIRS), large cerebral vessels such as middle cerebral artery (TCD), or in the arterioles and venules of the retina (DVA). Currently, there are limited data available on the simultaneous assessment of NVC responses using these methodologies.

Caffeine is the most commonly used stimulant drug with well documented effects on cerebral vasculature. Caffeine is known to non-specifically bind to adenosine receptors in the brain and to reduce resting blood flow while improving attention and cognitive function, which suggests that it may allow a more efficient dynamic blood flow regulation through neurovascular coupling. This study will use standardized dose of caffeine to test its effect on NVC responses in cerebral and retinal arterioles.

This study is designed to establish the direct link between reactivity in the cerebral and retinal micro- and macrovasculature. To achieve this goal, a prospective, single-blinded, placebo controlled, cross-over study will be employed to evaluate changes in the NVC responses measured simultaneously with DVA and TCD, or DVA and fNIRS before and after administration of 100mg of incapsulated caffeine or placebo pill.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Ability to read and write in English
* Competence to provide informed consent
* Non-occludable angle and with no optic neuropathy
* Subjects will be asked to refrain from caffeine consumption for at least 8 hours before participating in the study

Exclusion Criteria:

* The history of photosensitive epilepsy
* Intraocular pressure 21 Hgmm or higher
* Eyes with a visual acuity 20/30 or lower or the inability to fixate on fixation markers
* Previous symptoms of glaucoma attack (severe ocular pain and redness, decreased vision, colored halos in combination with headache, nausea and vomiting).
* Known allergies to study drugs
* Pregnancy and breast feeding
* Significant cardiac disease (e.g. heart failure), chest pain in the last 6 months
* Stage-2 high blood pressure not controlled by medication (>160/100 mm Hg)
* Uncontrolled diabetes mellitus; History of stroke; Multiple sclerosis; Chronic obstructive pulmonary disease; Active cancer; Abnormal liver function
* Diagnosis of dementia; Anxiety Disorder
* Absent temporal acoustic windows, intracranial stenosis (for TCD-related studies)
* History of arrhythmias
* Prisoners

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Modified Caffeine Research Visual Analogue Scales | Change from baseline measurements 1 hour after treatment
  Caffeine Research Visual Analogue Scales consists of seven visual analogue scales ("relaxed", "alert", "jittery", "tired", "tense", "headache", overall mood") are measured from 1 to 10 and have previously been used in research to evaluate the effects of caffeine. A single "mentally fatigued" visual analogue scale (scored from 1 to 10) will be included, as previous research has shown it to be sensitive to a caffeine-glucose drink.
Static retinal vessel assessment | Change from baseline measurements 1 hour after treatment
  Static analysis of retinal vasculature will be performed to evaluate averaged retinal arteriole and venule calibers. A ratio of these two measurements will be used to calculate arteriole-venule ratio.
Dynamic retinal vessel assessment | Change from baseline measurements 1 hour after treatment
  Flicker light-induced dilation of the retinal vessels (percentage increase over baseline diameter) will be measured in the right eye of each subject using the Dynamic Vessel Analyzer (DVA, IMEDOS Systems, Jena, Germany). The change in retinal vessel diameters is tracked and reported as a %change from baseline.
Cerebrovascular reactivity using transcranial Doppler | Change from baseline measurements 1 hour after treatment
  Transcranial Doppler sonography will be assessed simultaneously with the dynamic retinal vessel analysis and the blood flow velocity will be measured in the posterior cerebral artery. Change in the blood flow velocities from baseline will be measured.
Cerebrovascular reactivity using functional near infrared spectroscopy (fNIRS) | Change from baseline measurements 1 hour after treatment
  Functional near infrared spectroscopy (fNIRS) will be performed during the finger tapping task or go-no-go cognitive task. fNIRS approach generates data that represent a relative change in oxygenated and deoxygenated hemoglobin measured over the cortical brain tissues. Cerebrovascular reactivity will be evaluated as a change in oxy- and deoxy-hemoglobin between "during" and "before" task.

CONTACTS AND LOCATIONS:
Overall Officials: Andriy Yabluchanskiy, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Translational GeroScience Laboratory, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No